CLINICAL TRIAL: NCT05138133
Title: A Multicentre Randomized Double-Blind Placebo Controlled Phase 3 Study to Evaluate the Efficacy and Safety of Anifrolumab in Adult Patients With Active Proliferative Lupus Nephritis
Brief Title: Phase 3 Study of Anifrolumab in Adult Patients With Active Proliferative Lupus Nephritis
Acronym: IRIS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3466C00001; 2021-002862-42 (EudraCT Number)
Record Dates: First submitted 2021-11-17; First posted 2021-11-30 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Lupus Nephritis
Keywords: Lupus Nephritis, anifrolumab, Systemic Lupus Erythematosus, intravenous
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic | interventions — anifrolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind (Participant, Care Provider and Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Anifrolumab (Experimental): Solution for intravenous infusion
  Interventions: Drug: Anifrolumab
- Placebo (Placebo Comparator): Solution for intravenous infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anifrolumab — Anifrolumab intravenous infusion (IV)
  Other Names: Medi-546
  Arms: Anifrolumab
Drug: Placebo — Placebo intravenous infusion (IV)
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of IV antifrolumab in adult patients with Active Proliferative Lupus Nephritis

DETAILED DESCRIPTION:
This Phase 3, multicenter, multinational, randomized, double-blind, placebo-controlled study with OLE is to evaluate the efficacy and safety of anifrolumab versus placebo as added to SOC (MMF and glucocorticoids) in adults with active proliferative Class III or Class IV LN (both with or without concomitant Class V). The total study duration may be up to approximately 142 weeks, including screening and follow-up. Double-blind period will be 76 weeks. Participants who complete double-blind treatment period may enter open-label extension to receive anifrolumab for up 52 weeks. Approximately 360 of the enrolled participants will be randomly assigned to study intervention (anifrolumab or placebo) at a ratio of 1:1 during double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Active proliferative LN Class III or IV either with or without the presence of Class V according to the 2003 ISN/RPS classification
2. Renal biopsy obtained within 6 months prior to signing the ICF or during Screening Period.
3. Urine protein to creatinine ratio > 1 mg/mg (113.17 mg/mmol)
4. eGFR ≥ 35 mL/min/1.73 m2 (as calculated by the Chronic Kidney Disease Epidemiology Collaboration formula).
5. Fulfills updated 2019 EULAR/ACR SLE classification criteria.
6. No signs of symptoms of active TB prior to or during screening or no treatment for latent TB

Exclusion Criteria:

1. A diagnosis of pure Class V LN based on the renal biopsy obtained within 6 months prior to signing the ICF or during Screening.
2. Known history of a primary immunodeficiency, splenectomy, or any underlying condition that predisposes the participant to infection, or a positive result for HIV confirmed by the central lab at Screening - an HIV test must be performed during Screening, and the result should be available prior to Week 0 (Day 1).
3. Evidence of hepatitis C or active hepatitis B.
4. Any history of cancer except sucessfully cured skin squamos or basal skin carcinoma and cervical cancer in situ.
5. Receipt of the following for the current LN flare (ie, since the qualifying renal biopsy): IV cyclophosphamide > 2 pulses of high-dose (≥ 0.5 g/m2) or > 4 doses of low dose (500 mg every 2 weeks) or Average MMF > 2.5 g/day (or > 1800 mg/day of enteric coated mycophenolate sodium) for more than 8 weeks or Tacrolimus > 4 mg/day for more than 8 weeks; Cyclosporine for more than 8 weeks or during last 8 weeks prior to signing the ICF; Voclosporin for more than 8 weeks or during last 8 weeks prior to signing the ICF; Belimumab for more than 12 weeks or during last 12 weeks prior the ICF.
6. Previous receipt of >◦2 investigation treatments (other than anifrolumab) for LN or SLE since time of diagnosis and through the ICF.
7. Known intolerance to ≤ 1.0 g/day of MMF.
8. Any history of severe COVID-19 infection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2027-02-26 (Estimated); Study Completion 2028-12-05 (Estimated)

PRIMARY OUTCOMES:
Difference in proportion of participants with CRR (Complete Renal Response) in anifrolumab group compared with placebo group | Week 52
  CRR is defined as:
  * UPCR ≤ 0.5 mg/mg
  * eGFR ≥ 60 mL/min/1.73 m2 or no decrease from baseline of ≥ 20%

SECONDARY OUTCOMES:
Difference in proportion of participants achieving sustained OCS reduction in anifrolumab group compared with placebo group | from Week 24 through Week 52
  Sustained OCS reduction
HR of achieving sustained CRR in anifrolumab compared with placebo group | baseline through Week 52
  The endpoint for deriving the summary measure is time to sustained CRR, defined as time to achieving CRR that is sustained from that time point through week 52
Difference in the mean standardized AUC for UPCR between anifrolumab and placebo participants | baseline through Week 52
  Proteinuria as measured by the cumulative UPCR
Difference in proportion of participants with CRR in anifrolumab group compared with placebo group | Week 24
  CRR at week 24
HR to summarize the difference in the risk of hazard of renal-related event or death at any given time between anifrolumab and placebo participants | Through Week 52
  Onset of renal-related event or death through Week 52
HR to summarize the difference in the risk of hazard of renal-related event or death at any given time between anifrolumab and placebo participants | Through Week 76
  Onset of renal-related event or death through Week 76
Difference between anifrolumab and placebo in proportions of participants who achieve aCRR | Week 52
  aCRR (alternative complete renal response) defined as;
  * UPCR ≤ 0.5 mg/mg
  * eGFR ≥ 90 mL/min/1.73 m2 or no decrease from baseline of ≥ 10%
Difference between anifrolumab and placebo in proportions of participants who achieve CRR with sustained OCS reduction | Week 52
  CRR at Week 52 with Sustained OCS Reduction
HR of achieving sustained CRR in anifrolumab compared to placebo group | Through week 76
  Time to sustained CRR through the time frame period
HR of achieving 50% reduction in UPCR in anifrolumab compared to placebo group | Through Week 52
  The endpoint for deriving the summary measure is time from the first dose of study intervention to achieving 50% reduction in UPCR
Difference in mean UPCR between the anifrolumab and placebo group | Week 52
  Proteinuria as measured by UPCR
Difference in proportion of participants achieving PRR (Partial Renal Response) in anifrolumab group compared with placebo group | Week 52
  PRR defined as:
  UPCR <1.0 mg/mg (for participants with baseline UPCR ≤3 mg/mg) or >50% improvement and ≤3 mg/mg (for participants with baseline UPCR >3 mg/mg) eGFR
  ≥ 60 mL/min/1.73 m2 or no confirmed decrease of ≥20% from baseline
Difference in change from baseline in extra-renal SLEDAI-2K total score | Through Week 76
  The extra-renal SLEDAI-2K score is obtained by summing the SLEDAI-2K items without including the items within the renal system organ
Difference in mean change from baseline in domains and component scores of Short Form-36 Version 2 (SF-36v2) and Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-fatigue) total score | Week 52
  To evaluate patient-reported HRQOL and health status

CONTACTS AND LOCATIONS:
Locations (186):
- United States (31):
  - Research Site, Birmingham, Alabama
  - Research Site, Glendale, Arizona
  - Research Site, La Jolla, California
  - Research Site, La Palma, California
  - Research Site, Loma Linda, California
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, Upland, California
  - Research Site, New Haven, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Hallandale, Florida
  - Research Site, Plantation, Florida
  - Research Site, Sun City Center, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Louisville, Kentucky
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Newark, New Jersey
  - Research Site, Summit, New Jersey
  - Research Site, Las Cruces, New Mexico
  - Research Site, Great Neck, New York
  - Research Site, Manhasset, New York
  - Research Site, New York, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Middleburg Heights, Ohio
  - Research Site, Danville, Pennsylvania
  - Research Site, Allen, Texas
  - Research Site, Colleyville, Texas
  - Research Site, Edinburg, Texas
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
- Argentina (7):
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, La Plata
  - Research Site, Rosario
  - Research Site, San Juan
  - Research Site, San Miguel de Tucumán
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Leuven
  - Research Site, Liège
- Brazil (10):
  - Research Site, Belo Horizonte
  - Research Site, Campinas
  - Research Site, Cuiabá
  - Research Site, Juiz de Fora
  - Research Site, Maringá
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, Salvador
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Bulgaria (2):
  - Research Site, Plovdiv
  - Research Site, Sofia
- China (20):
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Jinan
  - Research Site, Jining
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Shanghai
  - Research Site, Shengyang
  - Research Site, Shenzhen
  - Research Site, Shijiazhuang
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Xi'an
  - Research Site, Zhengzhou
- Colombia (3):
  - Research Site, Barranquilla
  - Research Site, Cali
  - Research Site, Medellín
- France (6):
  - Research Site, Aurillac
  - Research Site, Bordeaux
  - Research Site, Marseille
  - Research Site, Paris
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Germany (9):
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Essen
  - Research Site, Göttingen
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Kirchheim
  - Research Site, Mainz Am Rhein
  - Research Site, Stuttgart
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Pécs
- India (12):
  - Research Site, Ahmedabad
  - Research Site, Dehradun
  - Research Site, Delhi
  - Research Site, Gurugram
  - Research Site, Hyderabad
  - Research Site, Kolkata
  - Research Site, Nadiād
  - Research Site, New Delhi
  - Research Site, Pune
  - Research Site, Secunderabad
  - Research Site, Vijayawada
  - Research Site, Visakapatnam
- Italy (8):
  - Research Site, Ancona
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Cona
  - Research Site, Eboli
  - Research Site, Monza
  - Research Site, Padua
  - Research Site, Roma
- Japan (20):
  - Research Site, Bunkyō City
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Gifu
  - Research Site, Hiroshima
  - Research Site, Izumo-shi
  - Research Site, Kita-gun
  - Research Site, Kitakyushu-shi
  - Research Site, Matsumoto-shi
  - Research Site, Nagasaki
  - Research Site, Okayama
  - Research Site, Ono
  - Research Site, Osaka
  - Research Site, Sagamihara-shi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shinagawa-ku
  - Research Site, Shinjuku-ku
  - Research Site, Toyoake-shi
- Malaysia (6):
  - Research Site, Batu Caves
  - Research Site, Ipoh
  - Research Site, Kajang
  - Research Site, Kuala Lumpur
  - Research Site, Kuantan
  - Research Site, Taiping
- Mexico (4):
  - Research Site, Chihuahua City
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, San Luis Potosí City
- Research Site, Amsterdam, Netherlands
- Peru (3):
  - Research Site, Bellavista
  - Research Site, Lima
  - Research Site, Piura
- Poland (10):
  - Research Site, Bydgoszcz
  - Research Site, Lodz
  - Research Site, Nadarzyn
  - Research Site, Olsztyn
  - Research Site, Opole
  - Research Site, Poznan
  - Research Site, Rzeszów
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Puerto Rico (2):
  - Research Site, Caguas
  - Research Site, San Juan
- Russia (6):
  - Research Site, Chelyabinsk
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Orenburg
  - Research Site, Saint Petersburg
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Hat Yai
  - Research Site, Muang
  - Research Site, Ratchathewi
- Turkey (Türkiye) (7):
  - Research Site, Adapazarı
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kahramanmaraş
  - Research Site, Kayseri
  - Research Site, Kocaeli
- Vietnam (4):
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean that all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Avasare R, Drexler Y, Caster DJ, Mitrofanova A, Jefferson JA. Management of Lupus Nephritis: New Treatments and Updated Guidelines. Kidney360. 2023 Oct 1;4(10):1503-1511. doi: 10.34067/KID.0000000000000230. PMID 37528520